CLINICAL TRIAL: NCT05374057
Title: Chiropractic Spinal Manipulative Therapy for Acute Neck Pain: a 4- Arm Clinical Placebo Randomized Controlled Trial
Brief Title: Chiropractic Spinal Manipulative Therapy for Acute Neck Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other); The Dam Foundation (Other)
Responsible Party: Principal Investigator, Michael Bjorn Russell, Project leader and co-supervisor, Professor of neurology, consultant neurologist, PhD, DrMedSci, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28498; 2021-005483-21 (EudraCT Number)
Record Dates: First submitted 2022-05-05; First posted 2022-05-13 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-03

CONDITIONS: Acute Neck Pain
Keywords: Randomized controlled trial (RCT); Clinical trial; Acute neck pain
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: A 4-arm parallel clinical placebo randomized controlled Trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants are blinded. The two chiropractor groups are single-blinded, while the two pharmacological groups are double-blinded. Chiropractor investigators are un-blinded in relation to the manual therapy they apply. Outcome assessors are blinded to group allocation of participants during the study and data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chiropractic Spinal Manipulative Therapy (CSMT) (Experimental): A specific contact, high-velocity, low-amplitude, spinal thrust manipulation directed to spinal biomechanical dysfunction in the cervical and/or thoracic spinal column, as diagnosed by standard chiropractic tests, in accordance with their clinical judgment.
  Interventions: Other: Chiropractic spinal manipulative therapy (CSMT)
- CSMT sham manipulation (Sham Comparator): A broad non-specific contact, low-velocity, low-amplitude sham push manoeuvre in a non-therapeutic directional line.
  Interventions: Other: CSMT sham manipulation
- Ibuprofen (Active Comparator): Ibuprofen 600mg, 3 times daily for 12 days.
  Interventions: Drug: Ibuprofen
- Placebo medication (Sham Comparator): Placebo medication, x 3 times daily for 12 days.
  Interventions: Drug: Placebo medication

INTERVENTIONS:
Other: Chiropractic spinal manipulative therapy (CSMT) — See study arm.
  Arms: Chiropractic Spinal Manipulative Therapy (CSMT)
Other: CSMT sham manipulation — See study arm.
  Arms: CSMT sham manipulation
Drug: Ibuprofen — See study arm.
  Other Names: Orifarm
  Arms: Ibuprofen
Drug: Placebo medication — See study arm.
  Other Names: Placebo
  Arms: Placebo medication

SUMMARY:
Acute neck is very common in the general population and often causes disability over shorter or longer time periods. Unfortunately, the efficacy of chiropractic spinal manipulative therapy (CSMT) and the efficacy of Non-steroidal Anti-inflammatory Drugs (NSAIDs) on acute neck pain is unknown. This 4-arm randomized controlled trial (RCT) will likely provide evidence for the efficacy of CSMT as well as NSAIDs. The applied methodology of the study will aim towards the highest research standards possible for manual-therapy RCTs, thus avoiding typical methodological shortcomings from previous manual-therapy studies. Our aim is to establish evidence-based knowledge on the efficacy of CSMT and NSAIDs in the treatment of acute neck pain.

DETAILED DESCRIPTION:
The Global Burden of Disease study ranks musculoskeletal neck pain as the most common disability worldwide. This study will highlight and validate CSMT for acute neck pain, compared to sham manipulation, ibuprofen and placebo medication. NSAIDs are the most frequently prescribed medications by GPs worldwide and are widely used for patients with back pain. However, evidence-based data are missing for acute neck pain patients treated with NSAIDs while existing evidence for CSMT for acute neck pain are limited by serious methodological shortcomings.

The 4-arm placebo-controlled RCT will assess the efficacy in the following four treatment groups:

1. Chiropractic spinal manipulative therapy (CSMT)
2. CSMT sham manipulation (placebo)
3. Ibuprofen (NSAID)
4. Placebo medication

We intend to invite 40 recruiting chiropractors from larger Norwegian cities, distributed by gender and geography. The study participants presenting to each chiropractor will be block-randomized equally into one of four study groups based on a computer-generated algorithm. Each chiropractor will include 16 participants, four into each arm. A total of 320 participants will be enrolled in the RCT, within 12 months. Participants randomized into the chiropractic treatment groups will receive 5 interventions over 12 days, i.e., CSMT or CSMT sham manipulation; while the pharmacological groups will receive 600mg ibuprofen or placebo administered 3 times daily for 12 days.

ELIGIBILITY:
Inclusion criteria

1. Eligible participants are between the age of 18 and 59 years old
2. Acute non-radicular neck pain, i.e., grade 1 or 2 according to the classification by the Bone and Joint Decade 2000-2010 Task Force on neck pain
3. Onset of the present episode ≤2 weeks prior to the 1st chiropractic visit
4. Moderate, severe or very severe pain intensity, i.e., ≥4, on a numeric rating scale (NRS) 0-10
5. Pain free for at least four consecutive weeks prior to the present pain episode
6. Not treated by a chiropractor during the past 3 months
7. Participants must accept not to seek other manual and/or pharmacological treatments for their acute neck pain during the intervention period
8. Non-pregnant women. Women in doubt shall have a negative fertility test before inclusion

Exclusion criteria

1. Contraindication to ibuprofen

   1. active peptic ulcer
   2. gastrointestinal bleeding
   3. previous repeated episode (≥2 detected events) with peptic ulcer or gastrointestinal bleeding
   4. previous gastrointestinal bleeding or ulcer using NSAIDs
   5. hypersensitivity to ibuprofen
   6. asthma induced by acetylsalicylic acid or other NSAIDs
   7. urticarial
   8. rhinitis
   9. severe heart failure (NYHA class IV)
   10. renal failure (glomerulus infusion <30 ml/min)
2. Taken pain- and/or anti-inflammatory medicine during the past 24 hours? (Patients that have taken acute pain- and/or anti-inflammatory medicine, including ibuprofen, can be included if they come back after 24 hours without having taken the medicine where they then fill out questionnaires and are randomized at the clinic)
3. On prescribed antidepressant
4. Major psychiatric disorder
5. Pregnancy or intention to be pregnant
6. Contraindication to SMT
7. Signs of spinal radiculopathy including progressive neurological deficit
8. Upper cervical spine instability (positive Sharp-Purser test)
9. Previous fracture in the cervical and/or thoracic spine
10. Previous cervical spine surgery
11. Recent (<6 months) severe physical trauma to the head, neck or thoracic spine within the previous 6 months
12. Concomitant low back pain with moderate, severe or very severe pain intensity (≥4 on a NRS)
13. Current chronic pain (defined as ≥3 months duration)
14. Rheumatoid arthritis
15. Recent (<2 weeks) acute respiratory infection with fever
16. Any presence of ischemic symptoms upon examination
17. Horner's syndrome
18. Medical history of arterial anomalies
19. History of connective tissue disorder
20. Familial history of cervical artery dissection
21. Other vascular disorders
22. Inability to understand instructions given in the Norwegian language
23. Inability to fill out digital questionnaires
24. Other reasons to exclude the patient as deemed necessary by the chiropractor

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Mean pain intensity change | From Day-0 to Day-14 between CSMT and sham CSMT, CSMT and ibuprofen, and CSMT and placebo medicine.
  Numerical Rating Scale (NRS) 0-10

SECONDARY OUTCOMES:
Mean pain intensity change | From Day-0 to Day-14. Comparison between ibuprofen and placebo medicine.
  Numerical Rating Scale (NRS) 0-10
Mean pain intensity change | From Day-0 to Day 2-13 in the treatment period, and from Day-0 to Day 7, 28, 56, 84 and 168 post-treatment, respectively, and comparison between CSMT and sham CSMT, CSMT and ibuprofen, CSMT and placebo medicine, ibuprofen and placebo medicine.
  Numerical Rating Scale (NRS) 0-10
Mean duration (hours) of neck pain change | From Day-0 to Day 2-13 and 14; From Day-0 to Day 7, 28, 56, 84 and 168 post-treatment, respectively, and comparison between CSMT and sham CSMT, CSMT and ibuprofen, CSMT and placebo medicine, ibuprofen and placebo medicine.
  Hours (0-24)
Mean number of days with neck pain per week | From the treatment period (14 days) to the periods; day 1-7, 22-28, 50-56, 78-84 and 162-168 post-treatment, respectively, and comparison between CSMT and sham CSMT, CSMT and ibuprofen, CSMT and placebo medicine, ibuprofen and placebo medicine.
  Weekly number of days
Proportions of participants with mean daily pain intensity reduction of ≥50%, ≥75% and 100% | From Day-0 to Day 2-13 and 14, and from Day-0 to Day 7, 28, 56, 84 and 168 post-treatment, respectively, and comparison between CSMT and sham CSMT, CSMT and ibuprofen, CSMT and placebo medicine, ibuprofen and placebo medicine.
  Numerical Rating Scale (NRS) 0-10
Proportions of participants with mean duration (hours) reduction of ≥50%, ≥75% and 100% | From Day-0 to Day 2-13 and 14, and from Day-0 to Day 7, 28, 56, 84 and 168 post-treatment, respectively, and comparison between CSMT and sham CSMT, CSMT and ibuprofen, CSMT and placebo medicine, ibuprofen and placebo medicine.
  Hours 0-24
Proportions of participants with mean reduction of number of days with neck pain per week of ≥50%, ≥75% and 100% | From the treatment period (14 days), to the periods: Day 1-7, 22-28, 50-56, 78-84 and 162-168 post-treatment, respectively, and comparison between CSMT and sham CSMT, CSMT and ibuprofen, CSMT and placebo medicine, ibuprofen and placebo medicine
  Weekly number of days
Improvement in Research and development 12 (RAND-12) score (12 questions each with 5 possible answers) | From Day-0 to Day-14, Day-84 and 168 post-treatment, respectively, comparison between CSMT and sham CSMT, CSMT and ibuprofen, CSMT and placebo medicine, ibuprofen and placebo medicine.
  RAND-12 Term Short Form Health Survey (0 to 100, with higher scores indicating better physical and mental health functioning)
Improvement in Neck Disability Index score (10 questions each with 6 possible answers) | From Day-0 to Day-14, Day-84 and 168 post-treatment, respectively, comparison between CSMT and sham CSMT, CSMT and ibuprofen, CSMT and placebo medicine, ibuprofen and placebo medicine.
  Neck Disability Index (0-100, where 0 = no disability and 100 = complete disability)
Adverse event (AE) analysis | Daily during intervention period (day 2-13). AE analysis of CSMT, sham CSMT, ibuprofen, and placebo medicine, and comparison between CSMT and sham CSMT, CSMT and ibuprofen, CSMT and placebo medicine, ibuprofen and placebo medicine.
  Within and between group adverse events analysis
Analysis of patients' blinding (Manual therapy) | Daily during intervention period (Day-0, Day 2-13). Analysis of CSMT and sham CSMT, and comparison between CSMT and sham CSMT.
  Numerical rating scale (NRS) 0-10 in relation to receiving real CSMT (0 absolutely unsure and 10 absolutely sure that real CSMT was received), irrespective of whether the patient received sham or real CSMT
Analysis of patients' blinding (Medicine) | Daily during intervention period (Day-0, Day 2-13). Analysis of ibuprofen and placebo medicine, and comparison between ibuprofen and placebo medicine.
  Numerical rating scale (NRS) 0-10 in relation to receiving ibuprofen (0 absolutely unsure and 10 absolutely sure that ibuprofen was received), irrespective of whether the patient received ibuprofen or placebo medicine
Patients' and chiropractors' expectations to treatment efficacy | Day-0
  Numerical rating scale (NRS) 0-10 (0 no expectation at all and 10 the highest possible expectation to treatment efficacy)
Analysis of patients' satisfaction to treatment efficacy | Day-14 of the intervention period
  Numerical rating scale (NRS) 0-10 (0 no satisfaction at all, and 10 the highest possible satisfaction)

OTHER OUTCOMES:
Sick leave | Mean number of days at Day-0 compared to Week-12 and Week-24 post-treatment.
  Number of days and grade of sick leave
Validation of user ID-number | All digital questionnaires from Day-0 to study completion, that is to 24-weeks follow-up.
  Number and proportions of incorrect typing of ID-numbers during digital questionnaire completion.
Facilitatory/inhibitory factors/dilemmas affecting recruitment Qualitative focus group interviews to explore facilitatory/inhibitory factors and possible dilemmas experienced by chiropractor investigators. | Up to 6 months
  Qualitative focus group interviews with all chiropractor investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. Russell, Professor, Study Director — Division for Research and Innovation, Akershus University Hospital, Norway; Aleksander Chaibi, PhD, Principal Investigator — Institute for Health and Society, Faculty of Medicine, University of Oslo, Norway
Locations (1):
- Michael B. Russell, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaibi A, Stavem K, Russell MB. Spinal Manipulative Therapy for Acute Neck Pain: A Systematic Review and Meta-Analysis of Randomised Controlled Trials. J Clin Med. 2021 Oct 28;10(21):5011. doi: 10.3390/jcm10215011. PMID 34768531
- [Background] Chaibi A, Saltyte Benth J, Bjorn Russell M. Validation of Placebo in a Manual Therapy Randomized Controlled Trial. Sci Rep. 2015 Jul 6;5:11774. doi: 10.1038/srep11774. PMID 26145718
- [Derived] Chaibi A, Allen-Unhammer A, Kopke Vollestad N, Russell MB. Chiropractic spinal manipulative therapy for acute neck pain: A 4-arm clinical placebo randomized controlled trial. A prospective study protocol. PLoS One. 2023 Dec 7;18(12):e0295115. doi: 10.1371/journal.pone.0295115. eCollection 2023. PMID 38060549
- See also: Background and rationale for the RCT — https://pubmed.ncbi.nlm.nih.gov/34768531/
- See also: CSMT Sham manipulation procedure — https://pubmed.ncbi.nlm.nih.gov/26145718/